CLINICAL TRIAL: NCT03323892
Title: Effect of Abstinence Duration on Embryo Development: a Prospective Sibling Oocyte Study
Brief Title: Effect of Abstinence Duration on Embryo Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Neelke De Munck, Clinical Embryologist, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017/271
Record Dates: First submitted 2017-09-05; First posted 2017-10-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Embryo Development
Keywords: preimplantation development; DNA fragmentation; abstinence duration

STUDY DESIGN:
Intervention Model Description: a prospective sibling oocyte study: both study arms will be applied to the oocytes of 1 patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 'normal' abstinence duration (Active Comparator): Patients follow the normal abstinence duration as asked by the physician (2-7 days). This sperm will be used to inject half of the oocytes Intervention = second sperm sample
  Interventions: Other: second masturbation
- short abstinence duration (Experimental): Patients will be asked to produce a second sperm sample, 2 hours after the first. This sperm will be used to inject the other half of the oocytes.
  Intervention = second sperm sample
  Interventions: Other: second masturbation

INTERVENTIONS:
Other: second masturbation — Husbands will be asked to produce a second sperm sample in the masturbatorium

SUMMARY:
The aim the investigators study is to analyze the embryo development if oocytes of the participants are injected with sperm from a longer or shorter (2 hours) abstinence duration.

DETAILED DESCRIPTION:
Participants undergoing an IVF treatment, are asked to respect an abstinence duration of 2-7 days. This is to obtain a sufficient number of motile sperm. A recent investigation, analyzed the quality (number and motility) of a sperm sample produced after an abstinence duration of 4 to 7 days, followed by a second sperm sample 2 hours later. The second sample (after 2 hours) was able to produce sperm cells with a higher motility. Not only has this short abstinence duration of 2 hours a positive effect on the motility, it will also reduce the sperm DNA damage, which again has a positive effect on embryo development. Because participants need gametes of high quality to obtain embryos with a high quality, the investigators want to investigate what the effect is of abstinence duration on embryo development.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for embryo development up to day 5
* at least 6 mature oocytes
* fresh ejaculates
* ICSI
* fresh embryo transfer or freeze all strategy
* all stimulation protocols
* concentration of >1x10^6 /ml sperm

Exclusion Criteria:

* IVF
* IVF versus ICSI patients
* chirurgical sperm
* acceptors of donor oocytes
* patients with PGD
* patients already enrolled in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Embryo development (blastocyst stage) | 1 year
  embryo development 5/6 of the preimplantation development
Embryo development (cleavage stage) | 1 year
  embryo development on day 3 of the preimplantation development

SECONDARY OUTCOMES:
Fertilization | 1 year
  number of fertilized oocytes per number of mature oocytes
Utilization rate | 1 year
  number of embryos used for transfer + cryopreserved for the patient
Sperm quality | 1 year
  concentration and motility
Sperm DNA fragmentation | 1 year
  analysis of non-viable sperm in the two samples
Clinical Pregnancies | 1 year
  pregnancies with a fetal heart beat

CONTACTS AND LOCATIONS:
Overall Officials: Neelke De Munck, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No
No data available for researchers others than the ones involved in the study